CLINICAL TRIAL: NCT04084470
Title: The Effects of the Different Bread Types of Fully Known Composition on Gastrointestinal Symptoms in Individuals With Non-coeliac Wheat Sensitivity.
Brief Title: Effects of Different Bread Types in NCWS
Acronym: BREAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University (Other)
Collaborators: Wageningen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: NL67466.068.18; METC18-032 (Other: METC azM/UM)
Record Dates: First submitted 2019-08-20; First posted 2019-09-10 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: Non-Coeliac Wheat Sensitivity (NCWS)
Keywords: Non-Coeliac Wheat Sensitivity; Wheat Sensitivity; Bread; Wheat; Gastrointestinal symptoms

STUDY DESIGN:
Intervention Model Description: Double-blind randomized cross-over study
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bread types 1, 2 and 3 (Active Comparator): Daily consumption of 5 slices of allocated bread type for three intervention days (separated by a wash-out period of at least 7 days).
  Interventions: Dietary Supplement: Different types of bread
- Bread types 4, 5 and 6 (Active Comparator): Daily consumption of 5 slices of allocated bread type for three intervention days (separated by a wash-out period of at least 7 days).
  Interventions: Dietary Supplement: Different types of bread

INTERVENTIONS:
Dietary Supplement: Different types of bread — Two studies comprising a double-blind randomized cross-over study. All subjects start with a run-in period of 3 days, thereafter they will receive three different types of bread in a randomized order for 1 day each, with a wash-out period of at least 7 days in between. Before test days 2 and 3, there is also a run-in period of three days.

SUMMARY:
Although wheat and gluten containing food products are generally considered to be healthy, a large number of individuals in the general population reduces or limits their intake and/or replaces wheat by other grains because of possible symptoms. This non-coeliac wheat sensitivity (NCWS) is accompanied by a range of (extra-)intestinal complaints soon after consuming wheat, which improve after wheat withdrawal. Evidence for a biological mechanism and for the exact contributing compound is limited. Furthermore, the impact of grain type, bread processing and the resulting compositional changes in bread on gastrointestinal tolerability in NCWS is unclear, especially as consumed part of a typical daily human diet.

The objective of this study is to investigate the effects of well-characterised breads on (extra-)intestinal symptoms in individuals with NWGS using two double-blind randomized cross-over design (study A and B). Subjects are required to avoid any products that cause GI symptoms (e.g. wheat products) during the trial. The investigators hypothesize that grain type and processing will have a different effect on the primary outcomes.

In addition, we want to explore the in vitro effect of each bread type on gut microbiota composition and activity.

ELIGIBILITY:
Inclusion Criteria:

* Develops of self-reported GI symptoms within 12 hours after a single intake of bread;
* Age between 18-70 years;
* Asymptomatic or only mildly symptomatic (overall) GI symptoms score with VAS < 30mm) while on the gluten-free/gluten-restricted diet;
* Must have a freezer (-18ºC) to store the study breads during the study;
* Willing and able to give written informed consent and to understand, participate and comply with the research project requirements.

Exclusion Criteria:

* Medical history of coeliac disease, wheat allergy, inflammatory bowel disease, presence of an organic gastrointestinal (GI) disease (such as inflammatory bowel disease) or other disease which may interfere with NCWS symptoms (upon judgment of the physician-clinical investigator (Dr. Keszthelyi, Gastroenterologist MUMC+));
* Previous major abdominal surgery or radiotherapy interfering with gastrointestinal function:

  * Uncomplicated appendectomy, cholecystectomy and hysterectomy allowed unless within the past 6 months;
  * Other surgery may be allowed based upon judgment of the physician-clinical investigator (Dr. Keszthelyi, Gastroenterologist MUMC+), who will decide on inor exclusion based upon the surgery applied;
* Use of medication potentially influencing gastrointestinal function and/or NCWS symptoms is allowed, provided that dosing has been stable for ≥ 1 month before enrolment;
* Administration of probiotic, prebiotic supplements, investigational drugs or participation in any scientific intervention study, which may interfere with this study (to be decided by the principle investigator), in the 14 days prior to the study;
* Excessive use of alcohol (>15 alcoholic units per week), or other drugs;
* Plan to lose weight or follow a specific weight loss diet within the study period;
* Current malignancy;
* Pregnancy or breastfeeding;
* Participation in any scientific intervention study, which may interfere with this study;
* Insufficient fluency of the Dutch language.

Follow-up measurement - inclusion criteria

* (1) NCWS subject: develops GI symptoms within 12 hours after consumption of at least one of the study breads of study A or B (+15 mm on VAS); OR (2) Healthy control (sex matched to NCWS subjects): eats bread regularly (min. 5 days per week)
* Age between 18-70 years;
* Must have a fridge (4-7ºC) to shortly store the collected faecal sample.

Follow-up measurement - exclusion criteria in addition to the criteria listed above:

* Use of antibiotics during the 6 past months prior to faecal sampling;
* Healthy controls: developing GI symptoms after consumption of bread, or following a gluten-free or wheat-free

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-09-17 (Actual); Primary Completion 2022-12-20 (Actual); Study Completion 2022-12-20 (Actual)

PRIMARY OUTCOMES:
Overall GI symptom score | At the end of day 1, 2 and 3 of the run-in period, at the end of test day 1, 2 and 3, and at the end of the last three days of each wash-out period (so the three days prior to testday 2 and 3).
  Change from baseline, measured on the Visual Analogue Scale ranged from 0 - 100, in which 0 is absence of symptoms and 100 is severe symptoms.

SECONDARY OUTCOMES:
Individual Intestinal symptom scores | At the end of day 1, 2 and 3 of the run-in period, at the end of test day 1, 2 and 3, and at the end of the last three days of each wash-out period (so the three days prior to testday 2 and 3).
  Change from baseline, measured on the Visual Analogue Scale ranged from 0 - 100, in which 0 is absence of symptoms and 100 is severe symptoms. Parameters: abdominal pain, abdominal discomfort, belching, bloating, flatulence, diarrhoea, constipation, urge to empty bowel, fullness, nausea.
Individual Extra-intestinal symptom scores | At the end of day 1, 2 and 3 of the run-in period, at the end of test day 1, 2 and 3, and at the end of the last three days of each wash-out period (so the three days prior to testday 2 and 3).
  Change from baseline, measured on the Visual Analogue Scale ranged from 0 - 100, in which 0 is absence of symptoms and 100 is severe symptoms. Parameters: tiredness, headache, joint pains, confusion, loss of coordination, skin rash.
Average stool frequency and consistency | After every stool production during day 1, 2 and 3 of the run-in period, during test day 1, 2 and 3, and during the last three days of each wash-out period (so the three days prior to testday 2 and 3).
  Bristol Stool Scale, a validated scale for faecal frequency and consistency, by classifying faeces into seven groups. Type 1: separate hard lumps, like nuts (hard to pass); Type 2: sausage-shaped but lumpy; Type 3: Like a sausage but with cracks on its surface; Type 4: Like a sausage or snake, smooth and soft; Type 5: Soft blobs with clear-cut edges (passed easily); Type 6: fluffy pieces with ragged edges, a mushy stool; Type 7: watery, no solid pieces / entirely liquid. Type 1-2 indicate constipation, type 3-4 are ideal stools as they are easier to pass, and type 5-7 may indicate diarrhoea and urgency.
Follow-up: microbiota composition | Follow-up measurement, within 1 year after completion of test day 3.
  After completion of the primary study, 5 responders (see in- and exclusion criteria) will be included for a follow-up measurement. For comparison, 5 healthy controls will be included. The participants will collect one fecal sample at home. These samples will be used to study the effect of the six different bread types on microbiota composition in an in vitro fermentation model.
Follow-up: microbiota activity | Follow-up measurement, within 1 year after completion of test day 3.
  After completion of the primary study, 5 responders (see in- and exclusion criteria) will be included for a follow-up measurement. For comparison, 5 healthy controls will be included. The participants will collect one fecal sample at home. These samples will be used to study the effect of the six different bread types on microbiota activity, measured by the release of microbial VOCs, in an in vitro fermentation model.

OTHER OUTCOMES:
Food intake by three-day food records | For 24 hours during day 1, 2 and 3 of the run-in period, during test day 1, 2 and 3, and during the last three days of each wash-out period (so the three days prior to test day 2 and 3).
  A three-day food record (on paper) to check for the adherence to the gluten-free diet.
Participant characteristics in relation to NCWS | Data on medical history and demographic factors will be collected during the screening visit as part of the screening process. Data on psychological factors will be collected after inclusion of subjects, before the start of the run-in period.
  To characterise NCWS subjects, data will be collected on medical history (e.g. surgery, GI diseases, medication use, allergies), demographic (e.g. age, gender, educational background, BMI, smoking, alcohol use) and psychosocial factors (relating to e.g. anxiety, depression, somatisation) using screening questionnaires.

CONTACTS AND LOCATIONS:
Overall Officials: Daisy MAE Jonkers, Prof., PhD, Principal Investigator — Maastricht University
Locations (2):
- Netherlands (2):
  - Maastricht University, Maastricht
  - Wageningen University, Wageningen

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] de Graaf MC, Timmers E, Bonekamp B, van Rooy G, Witteman BJ, Shewry PR, Lovegrove A, America AH, Gilissen LJ, Keszthelyi D, Brouns FJ, Jonkers DMAE. Two randomized crossover multicenter studies investigating gastrointestinal symptoms after bread consumption in individuals with noncoeliac wheat sensitivity: do wheat species and fermentation type matter? Am J Clin Nutr. 2024 Apr;119(4):896-907. doi: 10.1016/j.ajcnut.2024.02.008. Epub 2024 Feb 18. PMID 38373694